











## PARTICIPANT CONSENT FORM

**Study title:** Fetal Scalp Stimulation (FSS) versus Fetal Blood Sampling (FBS) to assess fetal wellbeing in labour – a multi-centre randomised controlled trial.

## Please initial the boxes

| I have read and understood the <b>Information Leaflet</b> about this study. The | Yes | No |
|---|---|---|
| information has been fully explained to me and I have been able to ask | | |
| questions, all of which have been answered to my satisfaction. | | |
| I understand that I don't have to take part in this study and that I can | Yes | No |
| withdraw at any time. I understand that I don't have to give a reason for my | | |
| withdrawal, and it won't affect my future medical care. | | |
| I am aware of the potential risks, benefits and alternatives of this research | Yes | No |
| study and consent to take part in the research. | | |
| I give permission for members of the research team in the Coombe and TCD | Yes | No |
| to look at my medical records to get information for this study. I have been | | |
| assured that information about me will be kept private and confidential. | | |
| I give permission for the Ethics Committee and any other representatives of | Yes | No |
| the Sponsor, or any regulatory authorities etc. to look at my baby's and my | | |
| medical notes to allow them to check that the study has been run safely. | | |
| I understand that the sponsor and Investigators have such insurance as is | Yes | No |
| required by law in the event of injury resulting from this research. | | |
| I have been given a copy of the Information Leaflet and this completed | Yes | No |
| consent form for my records. | | |
| I consent to take part in this research study having been fully informed of the | Yes | No |
| risks, benefits and alternatives. | | |
| I give informed explicit consent to have my data and my baby's data | Yes | No |
| processed as part of this research study. | | |
| I understand if I have any further questions, I can contact the Study Doctor | Yes | No |
| listed below. | | |
| I confirm that I have read and understood the UCC Data Protection Notice | Yes | No |
| that accompanied the Participant Information Leaflet | | |







| FUTURE CONTACT | | |
|---|---|---|
| I consent to be re-contacted by researchers about possible future research | Yes | No |
| related to the current study for which I may be eligible. | | |
| STORAGE AND FUTURE USE OF INFORMATION | \ | |
| I give permission for data to be stored for <i>possible future research related</i> | Yes | No |
| to the current study (fetal wellbeing in labour) without further consent being required but only if the research is approved by a Research Ethics | | |
| Committee. | | |
| Committee. | | |
| Name of Participant: | | |
| (Block Capitals) | | |
| (2.00m oup rous) | | |
| Signature of Participant: Date: Tim | e(24hr) | |
| To be assumed and by the Driverinal Investigator (Co. Investigator obtaining | | |
| To be completed by the Principal Investigator/Co-Investigator obtaining cons | sent. | |
| I, the undersigned, have taken the time to fully explain to the above patient th | e nature | and |
| purpose of this study in a way that they could understand. I have explained the | | |
| well as the possible benefits. I have invited them to ask questions on any aspe | | |
| that concerned them. | | , |
| Name (Block Capitals)Qualification: | | |
| Signature: Date: Time(24h | vr) | |
| Signature: Date: Time(24h | '' <i>/</i> | <del></del> |
| 3 copies to be made: 1 for participant, 1 for Study File and 1 for hospital media | al recor | ds. |